CLINICAL TRIAL: NCT04606888
Title: Transcutaneous Electrical Acupoint Stimulation for Postoperative Cognitive Dysfunction in Geriatric Patients With Gastrointestinal Tumor
Brief Title: Transcutaneous Electrical Acupoint Stimulation for Postoperative Cognitive Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Subei People's Hospital of Jiangsu Province (Other)
Responsible Party: Principal Investigator, Lijuan Xi, Principal Investigator, Subei People's Hospital of Jiangsu Province
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: LijuanXi
Record Dates: First submitted 2020-10-16; First posted 2020-10-28 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Postoperative Cognitive Dysfunction
Keywords: POCD; TEAS; Gastrointestinal tumor
MeSH Terms: conditions — Postoperative Cognitive Complications; Digestive System Neoplasms

STUDY DESIGN:
Intervention Model Description: Transcutaneous electrical acupoint stimulation group and control group
Who Masked: Participant, Outcomes Assessor
Masking Description: Patient don't konw which group they are in because we all told them that they will feel nothing during the intervention.
  The outcomes assessor just to evaluate indicators, they don't know the specific content of the patient's experiment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcutaneous electrical acupoint stimulation group (Experimental): Transcutaneous electrical acupoint stimulation group patients received Transcutaneous electrical acupoint stimulation (Neiguan [PC6], Yintang [GV 29], Zusanli [ST36]) for 30 min before the induction of anaesthesia until the end of the surgery and the night before operation, the first, second and third night after operation 30 min once a day with an altered frequency 2/100 Hz, disperse-dense waves, adjusted electricity intensity which was less than 10 mA.
  Interventions: Device: Transcutaneous electrical acupoint stimulation
- Control group (No Intervention): In Control group, except the electronic stimulation was not applied, the treatment was the same as the Transcutaneous electrical acupoint stimulation group.

INTERVENTIONS:
Device: Transcutaneous electrical acupoint stimulation — According to the traditional Chinese medicine 15,three acupuncture points were selected as the target points: bilateral Neiguan ,Yintang and bilateral Zusanli.. A transcutaneous electrical stimulator was used to provide an altered frequency 2/100 Hz,disperse-dense waves,and adjusted intensity which was less than 10mA.
  Arms: Transcutaneous electrical acupoint stimulation group

SUMMARY:
Postoperative cognitive dysfunction (POCD) is one of the common complications of cancer patients after operation with a 8.9%-46.1% incidence, which severely affecting patients' postoperative recovery, increasing the medical cost, affecting the social function of patients, reducing the quality of life and increasing the mortality.

Surgical trauma and perioperative pain can induce systematic inflammatory response and release systematic inflammatory mediators, which can enter the central nervous system (CNS) and lead to CNS inflammatory. In order to prevent the development of POCD among elder patients, the discovery of effective interventions reducing perioperative pain and inflammatory response is important.

Transcutaneous Electrical Acupoint Stimulation (TEAS) is a non-invasive alternative to needle-based electro-acupuncture (EA). It combines the acupuncture and transcutaneous electrical nerve stimulation (TENS) by pasting the electrode piece on the acupoint instead of sticking the needles on the skin. TEAS can trigger the release of endogenous neurotransmitters, releasing endogenous analgesic substances, such as endorphins. TEAS also can reduce the intraoperative anesthetic consumption, postoperative pain score, postoperative nausea and vomiting (PONV), and improve the postoperative recovery of patients. Recently, TEAS was found to improve the cognitive function of geriatric patients with silent lacunar infarction. However, the current TEAS mainly focus on intraoperative. The effect of perioperative TEAS on POCD is not clear.

Here, the effect of TEAS on POCD in geriatric adults undergoing radical resection of gastrointestinal tumors under general anesthesia was investigated to determine whether TEAS can decrease perioperative pain or inflammatory response to prevent the occurrence of POCD and to find out the relationship among perioperative TEAS, inflammatory response, postoperative pain, and POCD preliminarily.

DETAILED DESCRIPTION:
This study aims to evaluate the effect of perioperative transcutaneous electrical acupoint stimulation (TEAS) on postoperative cognitive dysfunction (POCD) in elderly patients who were diagnosed with gastrointestinal tumor and received radical resection of gastrointestinal tumors under general anesthesia and to determine the relationship among perioperative TEAS, inflammatory response, postoperative pain, and POCD preliminarily.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 60 years or older;
2. Patients were diagnosed with gastrointestinal tumor and received radical; resection of gastrointestinal tumors under general anesthesia in Subei people's hospital of Jiangsu province;
3. The patients understood the research content and signed the informed consent form;
4. American Society of Anesthesiology (ASA) score I-III;
5. No frailty before operation;
6. D-dimer was normal before the operation

Exclusion Criteria:

1. Patients with cognitive dysfunction before the operation or patients with previous history of cognitive dysfunction, dementia and delirium;
2. Patients with a history of severe depression, schizophrenia and other mental and nervous system diseases or taking antipsychotic or antidepressant drugs in the past;
3. Patients with severe hearing or visual impairment due to eye or ear diseases without assistive tools;
4. Patients who are unable to communicate or have difficulty communicating;
5. According to the definition of "China chronic disease and its risk factors monitoring report (2010)" (male average daily pure alcohol intake ≥ 61g, female average daily pure alcohol intake ≥ 41g, alcohol volume (g) = alcohol consumption (ML) × alcohol content% × 0.8);
6. Patients who were hospitalized for three months or more before surgery or who had received surgical treatment within three months;
7. Patients who can't take care of themselves or are physically disabled and unable to carry out nerve function test;
8. Patients with severe heart, liver and renal failure;
9. Patients with hypoxemia (blood oxygen saturation < 94%) more than 10 minutes during operation;
10. Patients admitted to ICU after operation;
11. Patients who quit or died due to noncooperation or sudden situation;
12. Patients who already participate in other clinical studies which may influence this study;
13. Patient who underwent emergency surgery;
14. Patient had a history of recent or conventional acupuncture treatment.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Mini-Mental State Examination score | In the morning of the day before operation
  Assess the cognitive function of the patient,the minimum value is 0,and the maximum value is 30, higher scores mean a better outcome.
Mini-Mental State Examination score | Three days after operation
  Assess the cognitive function of the patient,the minimum value is 0,and the maximum value is 30, higher scores mean a better outcome.
C reactive protein | The day before operation.
  Assess the inflammatory reaction of the patient
C reactive protein | The 1st day after the operation.
  Assess the inflammatory reaction of the patient
C reactive protein | The 3rd day after the operation.
  Assess the inflammatory reaction of the patient
Interleukin-6 | The day before operation.
  Assess the inflammatory reaction of the patient
Interleukin-6 | The 1st day after the operation.
  Assess the inflammatory reaction of the patient
Interleukin-6 | The 3rd day after the operation.
  Assess the inflammatory reaction of the patient
S100 calcium-binding protein β | The day before operation.
  Assess the inflammatory reaction of the patient
S100 calcium-binding protein β | The 1st day after the operation.
  Assess the inflammatory reaction of the patient
S100 calcium-binding protein β | The 3rd day after the operation.
  Assess the inflammatory reaction of the patient

SECONDARY OUTCOMES:
Numeric Rating Scale score | The day before operation
  Assess the pain score of the patient,the minimum value is 0,and the maximum value is 10, higher scores mean a worse outcome.
Numeric Rating Scale score | The day of operation
  Assess the pain score of the patient,the minimum value is 0,and the maximum value is 10, higher scores mean a worse outcome.
Numeric Rating Scale score | The 1st day after the operation.
  Assess the pain score of the patient,the minimum value is 0,and the maximum value is 10, higher scores mean a worse outcome.
Numeric Rating Scale score | The 2rd day after the operation.
  Assess the pain score of the patient,the minimum value is 0,and the maximum value is 10, higher scores mean a worse outcome.
Numeric Rating Scale score | The 3nd day after the operation.
  Assess the pain score of the patient,the minimum value is 0,and the maximum value is 10, higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Daorong Wang, Ph.D., Principal Investigator — Clinical Medical College of Yangzhou University
Locations (1):
- Northern Jiangsu People's Hospital, Yangzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
Underlie results in a publication
Supporting Information: Study Protocol
Time Frame: starting in October 2020
Access Criteria: Study which was used to do meta analyse

REFERENCES:
- [Background] Correction: Influence of postoperative analgesia on systemic inflammatory response and postoperative cognitive dysfunction after femoral fractures surgery: a randomized controlled trial. Reg Anesth Pain Med. 2019 Oct;44(10):e2. doi: 10.1136/rapm-2018-000023corr1. No abstract available. PMID 31534004
- [Background] Li Y, Huang D, Su D, Chen J, Yang L. Postoperative cognitive dysfunction after robot-assisted radical cystectomy (RARC) with cerebral oxygen monitoring an observational prospective cohort pilot study. BMC Anesthesiol. 2019 Nov 6;19(1):202. doi: 10.1186/s12871-019-0877-5. PMID 31694553
- [Background] Rasmussen LS, Johnson T, Kuipers HM, Kristensen D, Siersma VD, Vila P, Jolles J, Papaioannou A, Abildstrom H, Silverstein JH, Bonal JA, Raeder J, Nielsen IK, Korttila K, Munoz L, Dodds C, Hanning CD, Moller JT; ISPOCD2(International Study of Postoperative Cognitive Dysfunction) Investigators. Does anaesthesia cause postoperative cognitive dysfunction? A randomised study of regional versus general anaesthesia in 438 elderly patients. Acta Anaesthesiol Scand. 2003 Mar;47(3):260-6. doi: 10.1034/j.1399-6576.2003.00057.x. PMID 12648190
- [Background] Evered LA, Silbert BS. Postoperative Cognitive Dysfunction and Noncardiac Surgery. Anesth Analg. 2018 Aug;127(2):496-505. doi: 10.1213/ANE.0000000000003514. PMID 29889707
- [Background] Borges J, Moreira J, Moreira A, Santos A, Abelha FJ. [Impact of postoperative cognitive decline in quality of life: a prospective study]. Rev Bras Anestesiol. 2017 Jul-Aug;67(4):362-369. doi: 10.1016/j.bjan.2016.07.007. Epub 2017 Apr 12. Portuguese. PMID 28412051
- [Background] Kotekar N, Shenkar A, Nagaraj R. Postoperative cognitive dysfunction - current preventive strategies. Clin Interv Aging. 2018 Nov 8;13:2267-2273. doi: 10.2147/CIA.S133896. eCollection 2018. PMID 30519008
- [Background] Huang JM, Lv ZT, Zhang B, Jiang WX, Nie MB. Intravenous parecoxib for early postoperative cognitive dysfunction in elderly patients: evidence from a meta-analysis. Expert Rev Clin Pharmacol. 2020 Apr;13(4):451-460. doi: 10.1080/17512433.2020.1732815. Epub 2020 Feb 28. PMID 32077347
- [Background] Yang W, Kong LS, Zhu XX, Wang RX, Liu Y, Chen LR. Effect of dexmedetomidine on postoperative cognitive dysfunction and inflammation in patients after general anaesthesia: A PRISMA-compliant systematic review and meta-analysis. Medicine (Baltimore). 2019 May;98(18):e15383. doi: 10.1097/MD.0000000000015383. PMID 31045788
- [Background] Lv ZT, Huang JM, Zhang JM, Zhang JM, Guo JF, Chen AM. Effect of Ulinastatin in the Treatment of Postperative Cognitive Dysfunction: Review of Current Literature. Biomed Res Int. 2016;2016:2571080. doi: 10.1155/2016/2571080. Epub 2016 Aug 14. PMID 27597957
- [Background] Deng LQ, Hou LN, Song FX, Zhu HY, Zhao HY, Chen G, Li JJ. Effect of pre-emptive analgesia by continuous femoral nerve block on early postoperative cognitive function following total knee arthroplasty in elderly patients. Exp Ther Med. 2017 Apr;13(4):1592-1597. doi: 10.3892/etm.2017.4099. Epub 2017 Feb 3. PMID 28413514
- [Background] Zhang Q, Gao Z, Wang H, Ma L, Guo F, Zhong H, Xiong L, Wang Q. The effect of pre-treatment with transcutaneous electrical acupoint stimulation on the quality of recovery after ambulatory breast surgery: a prospective, randomised controlled trial. Anaesthesia. 2014 Aug;69(8):832-9. doi: 10.1111/anae.12639. Epub 2014 May 28. PMID 24865978
- [Background] Gao F, Zhang Q, Li Y, Tai Y, Xin X, Wang X, Wang Q. Transcutaneous electrical acupoint stimulation for prevention of postoperative delirium in geriatric patients with silent lacunar infarction: a preliminary study. Clin Interv Aging. 2018 Oct 24;13:2127-2134. doi: 10.2147/CIA.S183698. eCollection 2018. PMID 30425466
- [Derived] Xi L, Fang F, Yuan H, Wang D. Transcutaneous electrical acupoint stimulation for postoperative cognitive dysfunction in geriatric patients with gastrointestinal tumor: a randomized controlled trial. Trials. 2021 Aug 23;22(1):563. doi: 10.1186/s13063-021-05534-9. PMID 34425851